CLINICAL TRIAL: NCT01168804
Title: Bendamustine Plus Bortezomib Plus Dexamethasone in the Treatment of Stage II/III Relapsed or Refractory Multiple Myeloma
Brief Title: Bendamustine Plus Bortezomib Plus Dexamethasone in Relapsed or Refractory Multiple Myeloma
Acronym: BBD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Austrian Forum Against Cancer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBD
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; bendamustine; bortezomib; dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — Bendamustine Hydrochloride; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm bendamustine bortezomib dexamethasone (Experimental): single arm combination regimen: bendamustine - bortezomib- dexamethasone
  Interventions: Drug: bendamustine plus bortezomib plus dexamethasone

INTERVENTIONS:
Drug: bendamustine plus bortezomib plus dexamethasone — Bendamustine 70 mg/m2 on days 1+4 Velcade 1.3 mg/m2 on days 1,4,8,11 Dexamethasone 20 mg on days 1,4,8 and 11 Repeated every 4 weeks

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of the combination regimen of bortezomib-bendamustine-dexamethasone in patients with relapsed or refractory multiple myeloma

DETAILED DESCRIPTION:
After relapse after or early progression on first-line treatment the prognosis of multiple myeloma patients is unfavourable, with no remaining chance for cure. Therefore the search for new treatment regimens, including drugs with novel, and different, mechanisms of action is mandatory.

Both bendamustine and bortezomib are not yet established parts of standard first-line regimens, but showed to have high activity both in chemo-naïve and pre-treated patients. The novel mechanism of action of the proteasome inhibitor and the non-cross resistance of bendamustine to other alkylating agents established in the first-line treatment of multiple myeloma seem to recommend a combination of the two drugs for salvage therapy. The promising response data in a series of relapsing MM patients treated with bendamustine, bortezomib and prednisone support this assumption, as well as the feasibility and tolerability of the combination.

In summary, there is some evidence for a favourable risk/benefit ratio for the combination of bendamustine, bortezomib and a glucocorticoid drug, warranting the exploration in a larger, prospectively designed multicenter phase II study.

ELIGIBILITY:
Inclusion Criteria:

* Age min. 18 years at the time of signing the informed consent form
* Life expectancy of at least 3 months
* Able to adhere to the study visit schedule and other protocol requirements
* Measurable disease, defined as any quantifiable monoclonal protein value, defined by at least one of the following three measurements: Serum M-protein ≥ 10g/l; Urine light-chain (M-protein) of ≥ 200 mg/24 hours; Serum FLC assay: involved FLC level ≥10 mg/dl provided sFLC ratio is abnormal
* Relapsed or refractory MM in stage II or III after autologous SCT or conventional chemotherapy (histologically or cytologically proven/ Salmon and Durie criteria) in need of therapy
* All previous cancer therapy, including cytostatic therapy and surgery, must have been discontinued at least 4 weeks prior to treatment in this study, except corticosteroid therapy (dosage 40 to max. 160mg). Localised radiation therapy is allowed, but the increased risk of leukocytopenia, erythrocytopenia and thrombocytopenia based on the combination of a polychemotherapy and radiation therapy has to be considered and a close monitoring of the patients has to be assured.
* ECOG performance status of 0-2 at study entry
* Laboratory test results within these ranges:

  * Absolute neutrophil count min. 1.5 x 109/L
  * Platelet count min. 75 x 109/L
  * Total bilirubin max. 1.5 mg/dL
  * AST (SGOT) and ALT (SGPT) max. 2 x ULN or max. 5 x ULN if hepatic lesions are present.
* Disease free of prior malignancies for min. 5 years with exception of curatively treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast
* Fertile patients must use effective contraception during and for 6 months after study treatment

No study treatment or any other procedure within the framework of the trial (except for screening) will be performed in any patient prior to receipt of written informed consent.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Pregnant or breast feeding females
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Peripheral neuropathy or neuropathic pain of grade 2 or greater intensity, as defined by NCI CTCAE, version 3.0.
* Use of any other experimental drug or therapy within 28 days of pre-study visit.
* Known hypersensitivity to the study drugs
* Any prior use of bortezomib or bendamustine in the last six months
* Concurrent use of other anti-cancer agents or treatments other than those stated in this treatment plan
* Known positive for HIV or infectious hepatitis, type A, B or C
* Active, uncontrolled infections
* Acute diffuse infiltrative pulmonary disease and pericardial disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2010-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
efficacy | 8 cycles à 28 days plus follow-up phase
  evaluation of the overall response rate (sCR + CR + VGPR + PR + MR)

SECONDARY OUTCOMES:
efficacy and safety | 8 cycles à 28 days plus follow-up phase
  assessment of progression-free survival, overall survival, time to maximum response and toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Heinz P. Ludwig, Univ. Prof., Principal Investigator — Wilhelminenspital Vienna
Locations (8):
- Austria (7):
  - Medical University Hospital Graz, Graz
  - Hospital Elisabethinen Linz, Linz
  - LKH Salzburg, 3rd Med. Dept., Salzburg
  - Med. University Vienna, Clinic for Internal Medicine 1 (Hematology and Hemostaseology), Vienna
  - Hanusch Hospital Vienna, Vienna
  - Wilhelminenspital Vienna, Vienna
  - Clinic Wels-Grieskirchen, 4th Internal Dept., Wels
- Faculty Hospital Brno, Brno, Czechia

REFERENCES:
- See also: Related Info — http://www.onkologie.at